CLINICAL TRIAL: NCT06043999
Title: A Prospective, Multicenter, Randomized, Open, Parallel Controlled, Non-inferiority Clinical Trial of Salvage Chemoradiotherapy Versus Radical Total Mesorectal Excision in the Treatment of Intermediate-risk Early Middle-low Rectal Cancer After Local Resection
Brief Title: Salvage Chemotherapy Versus Total Mesorectal Resection for Local Resection Rectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIH-SCTVTMEFLR
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy Effect; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salvage adjuvant chemoradiotherapy group (Experimental): Patitents under local radical resection of rectal adenocarcinoma received:
  1. Concurrent adjuvant chemotherapy
  2. Adjuvant radiotherapy: long-course radiotherapy was planned in this study.
  Interventions: Other: Salavge Adjuvant Chemoradiotherapy
- Radical TME group (Active Comparator): Patitents under local radical resection of rectal adenocarcinoma received:
  Standard TME surgery was performed 3-4 weeks after local resection.
  Interventions: Procedure: Radical total mesorectal excision

INTERVENTIONS:
Procedure: Radical total mesorectal excision — Standard TME surgery was performed 3-4 weeks after local resection. The operation is roughly divided into the following steps:After abdominal exploration, gradually ligation and from the inferior mesenteric vessels, pay attention to protect the left ureter, reproductive blood vessels and upper abdominal nerve; The descending colon was fully mobilized and the splenic flexure was mobilized if necessary. Follow the principle of TME, perform sharp resection of the total mesorectum, and pay attention to the protection of the prostate, vagina, pelvic nerve, etc.For can be removed through double stapling technique in low former (LAR) need not inline sphincter resection (excluding cases), to must be inline sphincter resection can be turned to the anus operation (ditto), consistent way can choose according to the intraoperative situation drag anastomosis or manual suture or stapling anastomosis. Prophylactic loop colostomy of transverse colon or ileostomy is recommended.
  Arms: Radical TME group
Other: Salavge Adjuvant Chemoradiotherapy — Concurrent adjuvant chemotherapy:5-Fu or 5-Fu analogues based chemotherapy regimens were selected. CapeOx or capecitabine monotherapy or FOLFOX is recommended, and no more than 3 months.Adjuvant radiotherapy protocol:long-course radiotherapy protocol.a. Target definition: areas at high risk for recurrence of the primary tumor and regional lymphatic drainage.b. Radiotherapy technology: conventional radiotherapy, three-dimensional conformal radiotherapy, intensity modulated radiotherapy, image guided radiotherapy, etc.c. Radiation dose:DT of 45Gy,1.8Gy per fraction in 25 fractions, was recommended for the high-risk recurrence area of the primary tumor and the regional lymphatic drainage area.
  Arms: Salvage adjuvant chemoradiotherapy group

SUMMARY:
Whether to perform radical TME or salvage chemoradiotherapy after local resection of intermediate-risk T1 rectal cancer is still controversial. A study based on the National Cancer Data Center showed that, because of the need for organ preservation, rescue chemoradiotherapy after local resection of rectal cancer was used in 10% of patients with T1N0 tumors and in 40% of patients with T2N0 tumors. However, the local recurrence caused by non-TME surgery is still the focus of concern for clinicians and patients. Previous retrospective studies have shown that there is no significant difference in overall survival and disease free survival between salvage CRT group and salvage TME group for patients with early rectal cancer after local resection. Pathological pT2 after local resection is the only independent risk factor for disease-free survival. However, limited to a single center and small sample size, the recurrence caused by salvage radiotherapy and chemotherapy should still be alert. Given these concerns, there is an urgent need to identify a better treatment regimen that can ensure reliable oncologic outcomes after local resection. Therefore, with TME as the control group and salvage chemoradiotherapy as the experimental group, we conducted a prospective, randomized, multicenter, non-inferiority clinical trial of the treatment effect of patients with intermediate-risk T1 and clinical stage N0M0 rectal cancer after local resection, to provide high-level evidence-based medical evidence for the final choice of these two salvage treatment methods.

DETAILED DESCRIPTION:
In China, with the implementation of population-based early screening for colorectal cancer, more and more colorectal cancer are detected and diagnosed at an early stage. However, although operation method is improved, but it is reported that the radical rectal cancer surgery resection or by a combination of abdominal perineal resection (low) still has as much as 36% of surgical morbidity and functional prognosis and quality of life of the patients with a significant negative impact on. More than half of rectal cancer patients experienced different degrees of defecation disorder after surgery. Urinary incontinence, urinary retention and sexual dysfunction were also common. In addition, after total mesorectal excision (TME), patients often face many stoma-related complications such as stoma prolapse, bleeding, necrosis, and inability to reverse stoma. Dutch TME clinical studies reported ,19%of the patients with rectal cancer resection before low did not successfully complete protective colostomy HaiNa, long-term or permanent colostomy rate is as high as 40%. After abdominoperineal resection, up to 40% of patients develop perineal wound complications. Under the guidance of the previous concept of tumor control, the disadvantages caused by radical surgery seem to be acceptable. However, with the deepening of research, more and more scholars believe that early rectal cancer can be avoided by local resection to avoid the risk of postoperative disability caused by radical surgery.

However, neither the NCCN guidelines nor other widely used guidelines at home and abroad believe that local resection is safe only for low-risk Tl stage rectal cancer with good/intermediate differentiation and no lymphatic or vascular invasion, and the resection margin must be at least 1mm. Histological features associated with an increased risk of local recurrence include poor histological differentiation, deep submucosal invasion, lymphatic or vascular invasion, perineural invasion, SM3, and tumor size (pT1> 5cm). Under any high-risk histological characteristics, significantly increased the risk of lymph node metastasis after local excision, tumor prognosis is damaged, need total mesorectum excision. Step guide, colorectal cancer is achieved if the endoscopic cure, need to achieve without vascular/nerve invasion, high/medium differentiation, and no more than 1000(including m submucosal infiltration of such a request. However, JSPEN guidelines suggest that lymph node dissection is necessary for the two characteristics of tumor vertical resection margin and tumor budding. In 2016, Borstlap[et al. proposed a more detailed oncology classification for early rectal cancer for the first time, which separated rectal cancer patients with specific oncology characteristics from the traditional definition of high-risk rectal cancer. It found that patients with early-stage rectal cancer (pTl stage,3-5cm in diameter or less than 3cm with at least one high-risk factor; pT2 stage tumor diameter < 3cm and no high-risk factors) accounted for 75% of locally resected rectal cancers. But for such a high proportion of early in patients with rectal cancer, postoperative NCCN give advice is to choose the traditional adjuvant radiation and chemotherapy or remedial radical resection (chemoradiotherapy, CRT), stereotypes can abandon always shall choose the remedial radical remains to be seen, therefore, The salvage treatment of early rectal cancer classified as intermediate-risk needs further study.

Salvage chemoradiotherapy can achieve the purpose of organ preservation, and the quality of life of patients is significantly better than that of patients undergoing salvage surgery. A surface, based on the research of the national cancer data center T1N0 after local excision of rectal cancer patients with radiation and chemotherapy was 10%, and the T2 local excision of rectal cancer after chemoradiation is as high as 40%, partial resection of additional remedial chemoradiation contrast radical TME surgery three years DFS no statistical differences. However, the absence of lymph node dissection and radiation injury (such as radiation enteritis, perianal pain, etc.) do not make clinicians and patients completely prefer adjuvant chemoradiotherapy. In addition, due to the requirements of quality of life and anxiety of patients, doctors sometimes avoid completing total mesorectal resection (cTME) surgery for intermediate and high-risk tumors and turn to salvage chemoradiotherapy as an alternative. Clinical data to support this strategy are still lacking. As an alternative to organ preservation after local resection, whether adjuvant chemoradiotherapy can be a reliable salvage option remains controversial.

At present, there are great differences in the results of studies on salvage therapy for intermediate-risk rectal cancer patients after local resection. Most of these studies included patients with different local resection platforms and different baseline conditions such as age, gender, and T stage. The local recurrence rate of salvage chemoradiotherapy is as high as 14%, but the patients included in the studies are not strictly in the intermediate-risk group. In 2022, Lin Guole's team reported 110 patients with early rectal cancer who underwent local resection, and they were divided into CRT group and TME group according to the salvage treatment method selected. There was no significant difference in overall survival and disease-free survival between the two groups, and pathological stage pT2 after local resection was the only independent risk factor affecting disease-free survival. The treatment mode of local resection combined with salvage chemoradiotherapy has a good effect on the sexual function and anorectal function of patients. However, limited to a single center and a small sample size, the recurrence problem caused by salvage chemoradiotherapy should still be vigilant. Based on the above problems, we urgently need to ensure that dangerous risk early in patients with rectal cancer after partial resection of oncology result under the condition of reliable to determine a more optimal treatment, for this is a fairly high proportion of patients provide good clinical evidence to choose treatment, and we think, The identified "optimal solution" should strike an optimal balance between treatment-related complication rates and tumor control in early-stage rectal cancer.

In conclusion, we conducted a prospective, randomized, open, multicenter, parallel controlled, non-inferiority clinical trial of curative TME (control group) and salvage chemoradiotherapy (experimental group) in patients with intermediate risk T1 rectal cancer after local resection. This study can provide high-level evidence support for the final choice of these two salvage treatments for intermediate-risk early rectal cancer after local resection. In addition, it can also add a new layer to the personalized and precise treatment of rectal cancer, which will benefit more patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years;
2. Local radical resection of rectal adenocarcinoma (TEM, TAMIS, TSPM, EMR, ESD or polypectomy)
3. pT1 with a diameter of 3-5 cm, or a maximum diameter of 3 cm, and at least poor differentiation and/or lymphovascular invasion and/or perineural invasion and/or SM3;
4. The distance from the lower edge of the tumor to the anal verge was within 10cm on MRI at initial diagnosis;
5. clinical stage N0M0 at initial diagnosis;
6. no multiple colorectal cancer;
7. The heart, lung, liver and kidney function can tolerate surgery;
8. Patients and their families were able to understand and willing to participate in this study, and provided written informed consent

Exclusion Criteria:

1. complicated with other malignant tumors or a previous history of malignant tumors;
2. not suitable for subsequent chemoradiotherapy or surgery;
3. a history of inflammatory bowl disease (IBD) or familial adenomatous polyposis (FAP);
4. recently diagnosed with other malignant tumors;
5. ASA physical status ≥ IV and/or ECOG performance status > 2 points;
6. patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or combined with serious underlying diseases can not tolerate surgery;
7. a history of severe mental illness;
8. pregnant or lactating women;
9. Patients with other clinical or laboratory conditions were not considered to be eligible for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Three years disease-free survival rate | 3 years after intervention
  Disease-free survival was defined as the absence of clinical, radiologic, or pathological (consistent with the pathological type of the primary tumor) evidence of recurrence on systemic examination, colonoscopy, CT/MRI, PET-CT, or needle biopsy (if necessary)

SECONDARY OUTCOMES:
Three years local recurrence rate | 3 years after intervention
  Local tumor recurrence was defined as evidence of clinical, imaging, or pathological (consistent with the pathological type of the primary tumor) recurrence found in the pelvic region by digital rectal examination, colonoscopy, CT/MRI, PET-CT, or needle biopsy (if necessary)
Three years overall survival rate | 3 years after intervention
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Five years disease-free survival | 5 years after intervention
  Defined as the proportion of patients who did not experience any of the following events from the beginning of the randomized subgroup to the end of the third year, which included disease progression, local recurrence, distant metastasis, or second primary colorectal cancer, or death from any cause.
five years overall survival | 5 years after intervention
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Anal function | up to 24 weeks year after intervention
  wexner incontience score (0-20 0:poor 20:best)
sexual function | up to 24 weeks after intervention
  IIEF5 score evaluates erectile function in men {1-25noninterpretable score (score between 1 and 4), severe erectile dysfunction (score between 5 and 10), moderate erectile dysfunction (score between11 and 15）， mild erectile dysfunction (score between 16 and 20), and normal erectile function (score between 21 and25）}
EORTC QLQ-C30 | up to 24 weeks after intervention
  evalution quality of life (0-100 0:poor 100:best)
Urinary function | up to 24 weeks after intervention
  IPSS score assesses the urinary functional results in men (0-35 0:best 35: poor)

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wallner C, Lange MM, Bonsing BA, Maas CP, Wallace CN, Dabhoiwala NF, Rutten HJ, Lamers WH, Deruiter MC, van de Velde CJ; Cooperative Clinical Investigators of the Dutch Total Mesorectal Excision Trial. Causes of fecal and urinary incontinence after total mesorectal excision for rectal cancer based on cadaveric surgery: a study from the Cooperative Clinical Investigators of the Dutch total mesorectal excision trial. J Clin Oncol. 2008 Sep 20;26(27):4466-72. doi: 10.1200/JCO.2008.17.3062. PMID 18802159
- [Background] den Dulk M, Smit M, Peeters KC, Kranenbarg EM, Rutten HJ, Wiggers T, Putter H, van de Velde CJ; Dutch Colorectal Cancer Group. A multivariate analysis of limiting factors for stoma reversal in patients with rectal cancer entered into the total mesorectal excision (TME) trial: a retrospective study. Lancet Oncol. 2007 Apr;8(4):297-303. doi: 10.1016/S1470-2045(07)70047-5. PMID 17395102
- [Background] Marr R, Birbeck K, Garvican J, Macklin CP, Tiffin NJ, Parsons WJ, Dixon MF, Mapstone NP, Sebag-Montefiore D, Scott N, Johnston D, Sagar P, Finan P, Quirke P. The modern abdominoperineal excision: the next challenge after total mesorectal excision. Ann Surg. 2005 Jul;242(1):74-82. doi: 10.1097/01.sla.0000167926.60908.15. PMID 15973104
- [Background] Bach SP, Hill J, Monson JR, Simson JN, Lane L, Merrie A, Warren B, Mortensen NJ; Association of Coloproctology of Great Britain and Ireland Transanal Endoscopic Microsurgery (TEM) Collaboration. A predictive model for local recurrence after transanal endoscopic microsurgery for rectal cancer. Br J Surg. 2009 Mar;96(3):280-90. doi: 10.1002/bjs.6456. PMID 19224520
- [Background] Bosch SL, Teerenstra S, de Wilt JH, Cunningham C, Nagtegaal ID. Predicting lymph node metastasis in pT1 colorectal cancer: a systematic review of risk factors providing rationale for therapy decisions. Endoscopy. 2013 Oct;45(10):827-34. doi: 10.1055/s-0033-1344238. Epub 2013 Jul 24. PMID 23884793
- [Background] Diagnosis And Treatment Guidelines For Colorectal Cancer Working Group CSOCOC. Chinese Society of Clinical Oncology (CSCO) diagnosis and treatment guidelines for colorectal cancer 2018 (English version). Chin J Cancer Res. 2019 Feb;31(1):117-134. doi: 10.21147/j.issn.1000-9604.2019.01.07. No abstract available. PMID 30996570
- [Background] Hashiguchi Y, Muro K, Saito Y, Ito Y, Ajioka Y, Hamaguchi T, Hasegawa K, Hotta K, Ishida H, Ishiguro M, Ishihara S, Kanemitsu Y, Kinugasa Y, Murofushi K, Nakajima TE, Oka S, Tanaka T, Taniguchi H, Tsuji A, Uehara K, Ueno H, Yamanaka T, Yamazaki K, Yoshida M, Yoshino T, Itabashi M, Sakamaki K, Sano K, Shimada Y, Tanaka S, Uetake H, Yamaguchi S, Yamaguchi N, Kobayashi H, Matsuda K, Kotake K, Sugihara K; Japanese Society for Cancer of the Colon and Rectum. Japanese Society for Cancer of the Colon and Rectum (JSCCR) guidelines 2019 for the treatment of colorectal cancer. Int J Clin Oncol. 2020 Jan;25(1):1-42. doi: 10.1007/s10147-019-01485-z. Epub 2019 Jun 15. PMID 31203527
- [Background] Min BS, Kim NK, Ko YT, Lee KY, Baek SH, Cho CH, Sohn SK. Long-term oncologic results of patients with distal rectal cancer treated by local excision with or without adjuvant treatment. Int J Colorectal Dis. 2007 Nov;22(11):1325-30. doi: 10.1007/s00384-007-0339-2. Epub 2007 Jun 12. PMID 17571241
- [Background] Morino M, Allaix ME, Caldart M, Scozzari G, Arezzo A. Risk factors for recurrence after transanal endoscopic microsurgery for rectal malignant neoplasm. Surg Endosc. 2011 Nov;25(11):3683-90. doi: 10.1007/s00464-011-1777-z. Epub 2011 Jun 7. PMID 21647814
- [Background] Sun G, Tang Y, Li X, Meng J, Liang G. Analysis of 116 cases of rectal cancer treated by transanal local excision. World J Surg Oncol. 2014 Jul 9;12:202. doi: 10.1186/1477-7819-12-202. PMID 25008129
- [Background] Duek SD, Issa N, Hershko DD, Krausz MM. Outcome of transanal endoscopic microsurgery and adjuvant radiotherapy in patients with T2 rectal cancer. Dis Colon Rectum. 2008 Apr;51(4):379-84; discussion 384. doi: 10.1007/s10350-007-9164-5. Epub 2008 Jan 31. PMID 18236108
- [Background] Li Y, Qiu X, Shi W, Lin G. Adjuvant chemoradiotherapy versus radical surgery after transanal endoscopic microsurgery for intermediate pathological risk early rectal cancer: A single-center experience with long-term surveillance. Surgery. 2022 Apr;171(4):882-889. doi: 10.1016/j.surg.2021.08.044. Epub 2021 Oct 13. PMID 34656357